CLINICAL TRIAL: NCT00362739
Title: Collection of Blood for Gene Expression/Genomic Studies in Individuals With Chronic Lung Disease
Brief Title: Blood Collection From Individuals With Lung Disease for Genetic Studies
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0508008095
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Asthma; COPD; Interstitial Lung Disease; Cystic Fibrosis; Lung Cancer
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Cystic Fibrosis; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this study, a small amount of blood for extraction of DNA for the study of the genetic basis of lung disease will be obtained from each subject. The collected blood (cells and serum) will be used for genetic testing in studies relating to the genetic material and/or gene expression, and/or studies of proteins or other substances in serum (the liquid portion of the blood after it has been allowed to clot). Because these latter protein studies will occur at a future date, the serum will be stored for use in these studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Lung Disease: Individuals with at least one of the following: (1)symptoms consistent with pulmonary disease; (2) chest X-ray consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; (6) patients with diseases of organs with known association with lung disease; (7) individuals suspected of history of lung diseased based on history and/or physical examination
- 2: Normal Controls: Individuals without a history of lung disease

SUMMARY:
This is a research study where researchers are collecting blood to evaluate the genetic characteristics of individuals with chronic lung diseases, including asthma, chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, and lung cancer.

DETAILED DESCRIPTION:
The investigators hope to be able to identify an association between a genetic make-up in the blood samples and the risks of developing a particular lung disease, or severity of a lung disease. The findings of this study might be important to develop future preventative methods and potential treatments for the management of lung disease. The investigators aim to collect blood samples from 300 people with lung disease and 300 controls over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent
* Males and females, age 18 years and older
* Lung disease proven by at least one of the following:

  * symptoms consistent with pulmonary disease
  * chest X-rays consistent with lung disease
  * pulmonary function tests consistent with lung disease
  * lung biopsy consistent with lung disease
  * family history of lung disease
  * disease of organs with know associated with lung disease
  * individuals suspected of history of lung disease based on history and/or physical examination
  * normal controls (individuals without history of lung disease) to be sampled to provide a comparison to the lung disease cohort.

Exclusion Criteria:

* Drug and/or alcohol abuse within the past six months
* Females who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals visiting the Starr-5 Pulmonary, Critical Care Unit, and 5 West floor for standard clinical care will be recruited. Controls will be obtained from volunteers without a history of lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 3087 (Actual)
Dates: Start 2005-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Establish a set of normal ranges for various parameters in healthy individual specimens and compare to specimens from individuals with lung disease to determine parameters resulting in disease susceptibility and severity. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — The New York Presbyterian Hospital -- Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital -- Weill Cornell Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided